CLINICAL TRIAL: NCT07282834
Title: Randomized Phase II Trial of Heated Vs. Pressurized/Aerosolized Chemotherapy (HIPEC vs. PIPAC) for Peritoneal Carcinomatosis
Brief Title: Heated Versus Aerosol-based Laparoscopic Chemotherapy for Cancer That Has Spread to the Peritoneum (Abdominal Lining)
Acronym: Charlie-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Wagner, MD, FACS (Other)
Responsible Party: Sponsor-Investigator, Patrick Wagner, MD, FACS, Director, AHNCI Division of Complex General Surgical Oncology, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-177
Record Dates: First submitted 2025-10-30; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal (Metastatic) Cancer; Peritoneal Carcinomatosis; Abdominal Cancer; Abdominal Cancer Patients
Keywords: intraperitoneal; peritoneal cavity; mitomycin-C; PIPAC; HIPEC; Heated Intra-Peritoneal Chemotherapy; Pressurized Intraperitoneal Aerosol Chemotherapy; intra-abdominal; cytoreduction
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The treating investigator, participant and care provider will know which procedural arm the participant is assigned to after the enrollment visit has concluded and informed consent has been signed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heated Intra-Peritoneal Chemotherapy (HIPEC) Administration of Mitomycin C Chemotherapy (Active Comparator): Laparoscopic intraperitoneal administration of mitomycin C chemotherapy through peritoneal catheters, heated intra-peritoneal chemotherapy (HIPEC) delivered during surgical procedures.
  Interventions: Procedure: Heated intra-peritoneal chemotherapy
- Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Administration of Mitomycin C Chemotherapy (Active Comparator): Conventional administration of pressurized/aerosolized laparoscopic delivery of mitomycin C chemotherapy (PIPAC)
  Interventions: Procedure: Aerosolized intra-peritoneal chemotherapy

INTERVENTIONS:
Procedure: Heated intra-peritoneal chemotherapy — Mitomyocin C 40 mg will be administered in divided doses (30mg at time zero and 10mg at 60 minutes) for a total of 90 minutes at 41-43 degrees Celsius. Laparoscopic HIPEC will then be repeated laparoscopically up to two more times at 45 +/- 15 day intervals until three doses have been completed.
  Other Names: HIPEC
  Arms: Heated Intra-Peritoneal Chemotherapy (HIPEC) Administration of Mitomycin C Chemotherapy
Procedure: Aerosolized intra-peritoneal chemotherapy — PIPAC will be performed with mitomycin C, 12.5mg/m2, delivered laparoscopically for 30 minutes at ambient temperature. Laparoscopic PIPAC or be repeated laparoscopically up to two more times at 45 +/- 15 day intervals until three doses have been completed.
  Other Names: PIPAC
  Arms: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Administration of Mitomycin C Chemotherapy

SUMMARY:
This research study aims to improve the treatment of Peritoneal Carcinomatosis (PC), a condition where cancer spreads within the abdomen. Patients with PC often experience significant pain and nutritional problems. Currently, there isn't a standard treatment approach, and doctors use different combinations of chemotherapy, surgery, and methods to deliver chemotherapy directly into the abdomen (intra-peritoneal or "IP" chemotherapy).

The study will compare two IP chemotherapy methods: HIPEC and PIPAC. HIPEC involves circulating heated chemotherapy through the abdomen during surgery, while PIPAC delivers chemotherapy as a pressurized aerosol during a laparoscopic procedure. Both methods aim to achieve the same goal, but they haven't been directly compared to see which is safer, more tolerable, more effective, and provides better value.

DETAILED DESCRIPTION:
Mitomycin C is the chemotherapy that is being administered but it is not being evaluated in the study. Mitomycin C is an FDA-approved antineoplastic antibiotic, meaning it's a type of chemotherapy drug used to treat cancer. It works by interfering with DNA synthesis, which is essential for cell growth and division. By disrupting DNA, mitomycin C can prevent cancer cells from multiplying and spreading.

The study will enroll up to 200 patients who will be randomly assigned (like the flip of a coin) to receive either HIPEC or PIPAC. Participants will be active on the study for 120-180 days.

During the study, patients will undergo standard diagnostic laparoscopies (a minimally invasive surgical procedure) to assess their eligibility for surgery to remove as much cancer as possible. Before treatment begins, small tissue samples (biopsies) will be taken for analysis in the pathology department. A small portion of this tissue will be saved by the researchers to study the effects of treatment on tumors. Patients will then receive three rounds of chemotherapy administered by either HIPEC or PIPAC, each about six weeks apart, and each during a laparoscopic procedure. Tumor tissue biopsies will be collected at the time of each treatment for analysis in the pathology department, and a small portion of each biopsy will again be saved by the researchers for laboratory work to study the effects of the treatment on tumors.

Finally, patients will have another laparoscopy to assess the treatment's effect and check for any side effects. Although patients will be followed for up to 5 years, no study-specific follow-up visits are required. Participants undergoing this type of treatment also complete quality-of-life surveys at the start of the study, and after each IP chemotherapy treatment, that asks about general health, well-being and ability to do daily activities. Patient responses to these surveys are collected for research purposes.

HIPEC and PIPAC chemotherapy, are already standard ways to treat PC. This means there's no extra risk to study participants. However, as with any treatment, there are some potential risks, such as infection inside the abdomen or injury to organs during the procedure to deliver the chemotherapy. These risks are small and would be the same whether the participant were in the study or receiving these treatments as part of their normal care.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 to 80 years.
2. Biopsy-proven or clinically suspected peritoneal carcinomatosis
3. Receipt of at least three months of standard systemic chemotherapy prior with persistence of disease at the time of randomization
4. Not a candidate for surgical cytoreduction at the time of laparoscopy
5. Women at least 18 years of age of childbearing potential must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
6. Must be able to read and understand English and consent for themselves

Exclusion Criteria:

1. Patients who are eligible for definitive cytoreductive surgery at the time of enrollment
2. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease:

   AST/SGOT > 2.5 times the upper limit of normal ALT/SGPT > 2.5 times the upper limit of normal Total bilirubin > 2.5 times the upper limit of normal Hemoglobin < 7 gm/dL White blood cell count < 3,000/ mm3 Platelet count < 50,000/mm3
3. Any investigational drug use within 30 days prior to enrollment.
4. Systemic therapy within 14 days prior to randomization
5. Allergy or medical contra-indication to chemotherapy utilized in this study
6. Medical contraindication to laparoscopic surgery or complex cytoreductive surgery
7. Pregnant or lactating females.
8. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2040-11 (Estimated)

PRIMARY OUTCOMES:
Heated intra-peritoneal chemotherapy (HIPEC) Adverse Events | 150 days from Day #1 visit
  Frequency of drug-related adverse events following HIPEC as assessed by CTCAE v5
Heated intra-peritoneal chemotherapy (HIPEC) Surgical Complications | 150 days from Day #1 visit
  Frequency of surgical complications following HIPEC
Heated intra-peritoneal chemotherapy (HIPEC) Adverse Events | 150 days from Day #1 visit
  Severity of drug-related adverse events following HIPEC as assessed by CTCAE v5
Heated intra-peritoneal chemotherapy (HIPEC) Surgical Complications | 150 days from Day #1 visit
  Severity of surgical complications following HIPEC as assessed by using Clavien-Dindo scale
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Adverse Events | 150 days from Day #1 visit
  Frequency of drug-related adverse events following PIPAC as assessed by CTCAE v5
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Adverse Events | 150 days from Day #1 visit
  Severity of drug-related adverse events following PIPAC as assessed by CTCAE v5
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Surgical Complications | 150 days from Day #1 visit
  Frequency of surgical complications following PIPAC
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Surgical Complications | 150 days from Day #1 visit
  Severity of surgical complications as assessed following PIPAC by using Clavien-Dindo scale
Heated intra-peritoneal chemotherapy (HIPEC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of HIPEC as determined by length of hospital stay
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of PIPAC as determined by length of hospital stay
Heated intra-peritoneal chemotherapy (HIPEC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of HIPEC as determined by usage of pain medication in opioid equivalents prior to discharge
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of PIPAC as determined by usage of pain medication in opioid equivalents prior to discharge
Heated intra-peritoneal chemotherapy (HIPEC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of HIPEC as determined by patient-reported outcomes using the Short Form-20 instrument
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Tolerability | 150 days from Day #1 visit
  The relative tolerability of PIPAC as determined by patient-reported outcomes using the Short Form-20 instrument

SECONDARY OUTCOMES:
Heated Intra-Peritoneal Chemotherapy (HIPEC) Efficacy | 150 days from Day #1 visit
  Serological indicators of tumor response following HIPEC using serum levels of CEA, CA19-9 or CA-125 as applicable in individual patients
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Efficacy | 150 days from Day #1 visit
  Serological indicators of tumor response following PIPAC using serum levels of CEA, CA19-9 or CA-125 as applicable in individual patients
Heated Intra-Peritoneal Chemotherapy (HIPEC) Efficacy | 150 days from Day #1 visit
  Radiographic indicators of tumor response following HIPECusing RECIST criteria, when available.
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Efficacy | 150 days from Day #1 visit
  Radiographic indicators of tumor response following PIPAC using RECIST criteria, when available
Heated Intra-Peritoneal Chemotherapy (HIPEC) Efficacy | 5.5 years from Day #1 visit
  Proportion of patients achieving complete cytoreduction following HIPEC using the Completeness of Cytoreduction score
Pressurized Intraperitoneal Aerosol (PIPAC) Efficacy | 5.5 years from Day #1 visit
  Proportion of patients achieving complete cytoreduction following PIPAC using the Completeness of Cytoreduction score
Heated Intra-Peritoneal Chemotherapy (HIPEC) Efficacy | 5.5 years from Day #1 visit
  Total cost of care following PIPAC using hospital financial records to determine the total direct cost in US dollars
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Efficacy | 5.5 years from Day #1 visit
  Total cost of care following PIPAC using hospital financial records to determine the total direct cost in US dollars
Heated Intra-Peritoneal Chemotherapy (HIPEC) Efficacy | 150 days from Day #1 visit
  Biomarkers analysis of treatment response using tissue biopsy
Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) Efficacy | 150 days from Day #1 visit
  Biomarkers analysis of treatment response using tissue biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wagner, MD, Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny Health Network West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No